CLINICAL TRIAL: NCT03392220
Title: A Multicenter, Randomized, Case-control Study of Unilateral vs Bilateral Selective Neck Dissection for Clinically Negative Neck of Supraglottic Laryngeal Carcinoma
Brief Title: A Multicenter, Randomized, Case-control Study of Unilateral vs Bilateral Neck Dissection for cN0 Supraglottic Laryngeal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Hebei Medical University Fourth Hospital (Other); Jilin Provincial Tumor Hospital (Other); Jinzhou Medical University (Other)
Responsible Party: Principal Investigator, Wang Xiaolei, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-H&N-009
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Laryngeal Neoplasms; Malignant Neoplasm of Supraglottis Primary; Neck Dislocation
Keywords: clinically negative neck; regional control rate
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- undergo unilateral (affected side) neck dissection (II-IV) (Experimental): patient undergo affected side neck dissection, along with the excision of the laryngeal primary tumor
  Interventions: Procedure: Unilateral Neck Dissection
- undergo bilateral neck dissection (II-IV) (Experimental): patient undergo bilateral neck dissection, along with the excision of the laryngeal primary tumor
  Interventions: Procedure: Bilateral Neck Dissection

INTERVENTIONS:
Procedure: Unilateral Neck Dissection — patient undergo unilateral (affected side) neck dissection, along with the excision of the laryngeal primary tumor
  Arms: undergo unilateral (affected side) neck dissection (II-IV)
Procedure: Bilateral Neck Dissection — patient undergo bilateral neck dissection, along with the excision of the laryngeal primary tumor
  Arms: undergo bilateral neck dissection (II-IV)

SUMMARY:
Supraglottic laryngeal carcinoma patients with clinically negative neck (cN0) will be randomized divided into two groups. Patients in case group will undergo unilateral neck dissection (II-IV) while bilateral neck dissection (II-IV) in control group. Regional control rate is the primary endpoint and comparison will be made to see if unilateral dissection can get similar regional control as control group.

DETAILED DESCRIPTION:
Some retrospective analysises showed the low local recurrence rate of patients who accepted unilateral neck dissection with cN0 supraglottic laryngeal carcinoma. The aim of this study is to see if unilateral dissection can get similar regional control as bilateral dissection.

308 patients with cN0 supraglottic laryngeal carcinoma will be enrolled in five centers of northern China. Patients will be randomly assigned to 1: 1 ratio case group or control goup. Patients in case group will undergo unilateral (laryngeal primary tumor affected side) neck dissection (II-IV) while bilateral neck dissection (II-IV) in control group. And other necessary standard treatments will be performed in both case group and control group.Allowed by the patients, the investigators will obtain archived tumor specimens and 10ml peripheral blood samples from the patients before surgery.

The patients will be followed-up every three months after surgery, until three years after surgery or develop regional recurrence. During the follow-up procedure, radiological evaluation will be performed. The primary end point is the patient's pathologically confirmed regional lymph node recurrence. Patients with primary end point will enter the overall survival follow-up stage. At the median follow-up time of two years, the investigators will undergo a major regional control rate analysis, then, all patients will be followed-up to five years postoperatively, and the overall survival analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. The patients obtain informed consent prior to any trial.
2. Diagnosis: Histopathology was confirmed to be squamous cell carcinoma. Classified by laryngoscopy as supraglottic, no tongue and deep pharyngeal invasion, and subglottic invasion. Also, no distant signs of metastasis.
3. Primary lesion is limited to one side, violation or more than midline, but preoperative laryngoscopy and CT can still clearly distinguish between the severity of bilateral lesions.
4. Evaluation of cN0: Patients need to undergo neck palpation, ultrasound and enhanced CT, if the patient is allergic to CT enhancer, replace it with MRI.Not touch more than 2cm hard lymph nodes in the neck, moreover, ultrasound and enhanced CT are not found lymph node that diameter ≥ 1cm.Or, the size does not meet the above criteria, but find rim enhancement, central irregular or hypodensity, and with the surrounding tissue boundary is obscure, and other suspicious transfer signs.
5. After multidisciplinary discussion, the preferred treatment for patients is surgical treatment.
6. Patients with no other previous head and neck cancer, and neck did not receive radiation therapy, no deep neck surgery, skin resection excepted.

Exclusion Criteria:

1. Laryngeal carcinoma but not squamous cell carcinoma, or primary pathology includes non-squamous cell components.
2. Preoperative laryngoscopy assessment of primary lesions just in the middle or both sides of symmetry, can not distinguish which side is more serious.
3. No surgical indications, or initial treatment evaluation recommends non-surgical treatment.
4. The patient had other head and neck cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Local-regional control | 3 years
  The local-regional control time is defined as the time from the primary surgery to any confirmed local-regional(neck) lymph node metastasis. The metastasis should be confirmed by both image examination( ultra-sound/CT/MRI etc.) and pathology examination. The primary outcome measure is to compare the unilateral neck dissection group's local-regional control time with the bilateral neck dissection group. The local control benefit of the two groups is evaluated.

SECONDARY OUTCOMES:
Progression free survival, Overall survival | 5 years
  The progression free survival and the overall survival of the two groups of patients are being measured and compared with one and other, so the survival benefit of the two policy is evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolei Wang, MD, Principal Investigator — Cancer Hospital Chinese Academy of Medical Science
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Science, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No